CLINICAL TRIAL: NCT06580249
Title: Efficacy and Mechanism of Repetitive Transcranial Magnetic Stimulation on the Symptoms of Pleasure Deficit in Adolescent Depression
Brief Title: Efficacy and Mechanism of rTMS on the Symptoms of Pleasure Deficit in Adolescent Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242219-C-1
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: pleasure deficit; repetitive transcranial magnetic stimulation; adolescent
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive transcranial magnetic stimulation true stimulation and sertraline treatment (Experimental): The rTMS was administered once a day, implementing approximately 10-20 minutes of physical therapy, with stimulation parameters of 10 Hz frequency, 120% MT intensity, and 50 treatment sequences of 60 stimulations each, with 30-second intervals between the sequences, for a total of 3000 stimulations. For medication: If the depressive episode is only monophasic, give sertraline hydrochloride tablets 1-2 tablets/day for treatment； if the patient has bipolar disorder-depressive episode, give the emotion stabilizer lithium carbonate tablets 0.5-1.0 g/day (adjust the dose according to the blood concentration) for treatment.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham Repetitive transcranial magnetic stimulation stimulation + sertraline treatment group (Sham Comparator): Pseudo stimulation mimicked the tactile and acoustic sensations of rTMS by flipping the head, at 90 degrees to the scalp, with other intervention parameters remaining consistent with the study group. For medication: If the depressive episode is only monophasic, give sertraline hydrochloride tablets 1-2 tablets/day for treatment； if the patient has bipolar disorder-depressive episode, give the emotion stabilizer lithium carbonate tablets 0.5-1.0 g/day (adjust the dose according to the blood concentration) for treatment.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — The true stimulus group acted directly, whereas the pseudo stimulus group reversed the head to produce no effect. Both groups were treated with sertraline medication。

SUMMARY:
(1) Primary objective: to collect data on the score of pleasure deficit scale before and after repetitive transcranial magnetic stimulation treatment in adolescent depressed patients, and to verify its efficacy and safety in adolescent depressed patients in combination with the changes of clinical symptoms; (2) Secondary objective: to explore the relevant hemodynamic mechanisms in adolescent depressed patients before and after repetitive transcranial magnetic stimulation treatment.

DETAILED DESCRIPTION:
Depression is one of the most common mental disorders among adolescents and is characterized by persistent low mood. According to a global statistical report released by the World Health Organization, about 350 million people worldwide are affected by depression, with the adolescent population being particularly prominent. Epidemiologic surveys in the Chinese region show that the prevalence of depression in adolescents is about 3.0%. The study points out that age is one of the key factors affecting major depression. Pleasure deficit, a reduced capacity for the experience of pleasure or a lack of appropriate emotional responses to rewards and positive stimuli, is a core symptom of depression and is considered a key internal phenotype of the illness. Repetitive transcranial magnetic stimulation is a treatment for major depressive disorder that delivers a series of equally spaced pulses through repetitive TMS. Studies have shown that rTMS stimulation of the dorsolateral prefrontal cortex can significantly improve symptoms of pleasure deficit. Thus, rTMS may be an effective treatment option for depressed patients with pleasure deficit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-19 years old (both 10 and 19), gender is not limited;
2. Meet the criteria for diagnosing MDD in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
3. First episode or relapse, monophasic or bipolar depressive disorder;
4. No history of any form of antidepressant treatment (including medication, physical and psychotherapy) within 2 weeks prior to enrollment;
5. Habitual right-handedness;
6. Deficit of pleasure scale (DARS) <22 points;
7. Score >17 on the 17-item version of the Hamilton Depression Scale (HAMD-17);
8. After fully understanding the safety of rTMS, they were willing to actively cooperate with the treatment and signed an informed consent form.

Exclusion Criteria:

1. Complicated with psychotic symptoms;
2. Comorbidity with major psychiatric disorders such as schizophrenia, delusional disorder, delirium, neurocognitive disorder, intellectual disability, and other mental disorders caused by other diseases;
3. History of primary neurologic disease or brain injury;
4. History of electroconvulsive therapy;
5. Contraindications to rTMS treatment, including cardiac pacemakers, neurostimulators, artificial metal heart valves, intracranial aneurysm clips, cochlear implants, and other types of metal implants (with the exception of oral supports);(6)History of epilepsy.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Difference in Scores on the Dimensional Anhedonia Rating Scale (DARS) in Patients from Baseline to 8 Weeks Post-Treatment | at baseline, at the end of treatment on day 7, at the end of treatment on day 14, 4 weeks after treatment, and 8 weeks after treatment
  The Dimensional Anhedonia Rating Scale, a relatively new tool for assessing symptoms of pleasure deficit, is a self-rating scale. It consists of four sections and 17 questions that focus on the patient's experience of pleasure in the present moment. Each question is rated on a 5-point scale of 1 (never), 2 (occasionally), 3 (sometimes), 4 (often), and 5 (always).The lower the DARS score, the greater the degree of pleasure deficit.

SECONDARY OUTCOMES:
Change in Difference in Scores of Patients' HAMD-17 Scores from Baseline to 8 Weeks Post-Treatment | at baseline, at the end of treatment on day 7, at the end of treatment on day 14, 4 weeks after treatment, and 8 weeks after treatment
  The Hamilton Depression Scale has 17 entries, each of which is categorized into either 5 levels or 3 levels. The scale has a minimum score of zero and a maximum score ranging from 2 to 4 for each rating item. The higher the patient's score, the more severe the depression.
Change in Difference in Scores on the Snaith-Hamilton Pleasure Scale (SHAPS) in Patients from Baseline to 8 Weeks Post-Treatment | at baseline, at the end of treatment on day 7, at the end of treatment on day 14, 4 weeks after treatment, and 8 weeks after treatment
  The Snaith-Hamilton Pleasure Scale has 14 entries, each of which is categorized into 4 levels. The scale has a maximum score of 56 and a minimum score of up to 14. The higher the patient's score, the more severe the pleasure deficit.
Change in Difference in Patient Temporal Experience of Pleasure Scale (TEPS) Scores from Baseline to 8 Weeks Post-Treatment | at baseline, at the end of treatment on day 7, at the end of treatment on day 14, 4 weeks after treatment, and 8 weeks after treatment
  The Temporal Experience of Pleasure Scale has 20 entries, each of which is categorized into 6 levels. The scale has a minimum score of 1 and a maximum score of 6 for each rating item. The lower the patient's score, the more severe the pleasure deficit.
functional near-infrared spectroscopy tests were performed from baseline to the end of week 2 of treatment. | at baseline, at the end of treatment on day 14
  Before and after treatment, near-infrared functional brain imaging was performed on each patient to monitor blood oxygen levels in each brain region and ultimately to compare hemodynamic changes before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- XijingH, Xi'an, Shaanxi, China